CLINICAL TRIAL: NCT03140774
Title: Evaluating the Long Term Immunogenicity of Ebola Virus Vaccines Ad26-ZEBOV, MVA-BN-Filo and rVSV-ZEBOV
Brief Title: Persistence of the Immune Response After Immunisation With Ebola Virus Vaccines
Acronym: PRISM
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: OVG2016/04
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2019-12

CONDITIONS: Ebola Virus Disease
Keywords: Ebola vaccine; immunogenicity; persistence
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will seek consent for storage of excess blood samples in the Biobank. Participants will be separately consented for this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Phase 1 participants: Previously exposed to Ebola vaccine Ad26-ZEBOV and MVA-BN-Filo.
  Interventions: Biological: Previously exposed to Ebola vaccine
- Cohort 2: Received r-VSV-ZEBOV vaccine: Previously exposed to Ebola vaccine rVSV-EBOV.
  Interventions: Biological: Previously exposed to Ebola vaccine
- Cohort 3: Phase 2 participants: Previously exposed to Ebola vaccine Ad26-ZEBOV and MVA-BN-Filo
  Interventions: Biological: Previously exposed to Ebola vaccine

INTERVENTIONS:
Biological: Previously exposed to Ebola vaccine — Exposure of interest: participants must have had one or more previous Ebola vaccines, Ad26.ZEBOV , MVA-BN-Filo or r-VSV-ZEBOV to enter the study.

SUMMARY:
The aim of this study is to investigate the persistence of the vaccine induced immune response between 24 - 60 months following primary vaccination.

The study consists of three cohorts:

Cohort 1: volunteers from the Phase 1 study of the various prime/boost regimes with two viral vectored Ebola vaccines: Ad26-ZEBOV and MVA-BN-Filo vaccines

Cohort 2: volunteers who have been vaccinated previously with Ebola vaccine r-VSV-ZEBOV

Cohort 3: volunteers from the Phase 2 study of 3 prime/boost regimes with Ad26.ZEBOV and MVA-BN-Filo vaccines (VAC52150EBL2001: EVOLVE).

DETAILED DESCRIPTION:
The Ebola Virus Disease (EVD), is caused by the viruses belonging to the genus Ebola virus. The disease occurs in sporadic outbreaks in the endemic zones of Africa and results in high mortality. During an outbreak, human to human to transmission occurs by contact with the body fluids of an infected individual. In the inter-endemic period the disease is zoonotically sustained in the environment. Prevention or control of future endemic outbreaks in the high risk areas of Africa will require effective preventative strategies including immunisation.

Cohort 1:

The Phase 1 study with the multiple heterologous prime boost regimes of the Ad26-ZEBOV and the MVA-BN-Filo vaccines demonstrated a substantive immunogenicity and safety of the vaccines. A combined immune response of humoral and cellular immunity was observed in the study participants. Furthermore, persistence of the immune response was evident at one year following the primary vaccination. It is not known whether the immune response persists beyond this time point. The duration of the immunological response is important as it will inform the clinical utility of the vaccines and whether or not additional booster dosage will be required and if so, at what interval.

In this study we will invite the 56 participants from the Phase 1 study at two time points: 24 - 30 months and 36 - 48 months after receiving the primary vaccination. Following consenting and enrolment into the study, the participants will undergo a blood test. We will assess the humoral immunity by estimating the level of binding antibody to the Ebola virus envelope glycoprotein. Cellular immunity will be assessed by estimating the functional CD4+ and the CD8+ T cells secreting the pro-inflammatory cytokines. We will undertake this assessment by intracellular staining of the peripheral blood mononuclear cells (PBMC) and using flowcytometry technique to identify the positively stained cells. A second assessment of the cellular immunity will be carried out by an in-house ELISpot technique subject to availability of additional funding.

Cohort 2:

In October 2015, contacts of a laboratory-confirmed case of Ebola virus diseases (EVD) in the U.K. were given the rVSV-EBOV vaccine as a part of clinical preventative care. Subsequently, these recipients of the rVSV-EBOV vaccine were enrolled and followed up for safety and immune response until one year post vaccination in the Glasgow Ebola Vaccine Follow-up Study (REC reference 15/WS/0251). The duration of persistence of the immune response to rVSV-EBOV beyond 360 days is unknown and may impact on the use of the vaccine in any future Ebola outbreaks. This study provides an opportunity to study the immune response beyond 1 year from the prime vaccination and to compare those results with the response to MVA-BN-Filo and Ad26-ZEBOV vaccines. This study will also allow for a further period of safety follow-up for this cohort.

Twenty-six individuals were vaccinated with the r-VSV-EBOV Ebola vaccine in Glasgow following possible exposure to a patient with confirmed Ebola virus disease as a part of preventative clinical care. All 26 individuals will be invited to take part in this study.

Cohort 3:

This cohort consists of participants from the Phase 2 study of 3 prime/boost regimes with Ad26.ZEBOV and MVA-BN-Filo vaccines (VAC52150EBL2001: EVOLVE). This was a randomized, observer-blind, placebo-controlled, parallel-group, multicentre, Phase 2 study to evaluate the safety, tolerability and immunogenicity of 3 heterologous prime-boost regimens which differed in the timing of the boost vaccination. The dose of each study vaccine (Ad26.ZEBOV, MVA-BN-Filo or placebo) and the sequence of vaccination were identical in each group. The prime/boost regimens were commenced in July 2015 and completed in February 2016.

Recruitment of participants in Group 1 (unblinded) of EVOLVE into the PRISM study can commence once all approvals are in place. However, for participants in Group 2 (blinded) of the EVOLVE study, recruitment and enrolment will not commence until after EVOLVE has been unblinded (anticipated to occur in Q4 2018 - Q1 2019).

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study.
2. Aged 18 years or above.
3. Subject must have received both vaccines in the phase 1 trial (Cohort 1) the r-VSV-ZEBOV vaccine (Cohort 2), or both vaccines in the Phase 2 trial (Cohort 3)
4. Agree to allow his or her General Practitioner and or Consultant if appropriate, to be notified of participation in the study, if required.

Exclusion Criteria:

1. History of malignancy and receipt of immunosuppressive therapy
2. Post organ or stem cell transplantation with or without follow-on immunosuppressive therapy
3. Receipt of adeno virus or MVA virus based vaccine since the Phase 1 or Phase 2 study (Cohort 1 and 3) or since receiving the r-VSV-ZEBOV vaccine (Cohort 2)
4. Chronic or recurrent use of medication which modify host immune response
5. A visit to an Ebola endemic area since the Phase 1 or Phase 2 study (Cohort 1 and 3) or since receiving the r-VSV-ZEBOV vaccine (Cohort 2)
6. Any contraindication to venepuncture, as determined by clinical judgement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1: 56 Phase 1 study participants who have received both Ad26-ZEBOV and the MVA-BN-Filo vaccines and who meet the inclusion and exclusion criteria as listed above .
  Cohort 2: 26 participants who received r-VSV-ZEBOV vaccine as a part of clinical preventative care.
  Cohort 3: 148 Phase 2 study participants who have received both Ad26-ZEBOV and the MVA-BN-Filo vaccines and who meet the inclusion and exclusion criteria as listed above
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Humoral Immunity | 24 to 60 months following the primary vaccination
  Binding antibody to the Ebola viral glycoprotein (GP) antigen assessed by ELISA

SECONDARY OUTCOMES:
Cellular Immunity | 24 to 60 months following the primary vaccination
  Pro-inflammatory cytokine response of T cells, by using intracellular staining technique and multicolour flow cytometer

OTHER OUTCOMES:
Cellular Immunity by alternative method | 24 to 60 months following the primary vaccination
  Interferon-gamma (INF-gamma) release by Ebola GP specific activated T cells as measured by ELISpot

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Snape, FRCPH, MD, Principal Investigator — Oxford Vaccine Group, University of Oxford
Locations (2):
- United Kingdom (2):
  - MRC - University of Glasgow Centre for Virus Research, Glasgow
  - Oxford Vaccine Group, University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milligan ID, Gibani MM, Sewell R, Clutterbuck EA, Campbell D, Plested E, Nuthall E, Voysey M, Silva-Reyes L, McElrath MJ, De Rosa SC, Frahm N, Cohen KW, Shukarev G, Orzabal N, van Duijnhoven W, Truyers C, Bachmayer N, Splinter D, Samy N, Pau MG, Schuitemaker H, Luhn K, Callendret B, Van Hoof J, Douoguih M, Ewer K, Angus B, Pollard AJ, Snape MD. Safety and Immunogenicity of Novel Adenovirus Type 26- and Modified Vaccinia Ankara-Vectored Ebola Vaccines: A Randomized Clinical Trial. JAMA. 2016 Apr 19;315(15):1610-23. doi: 10.1001/jama.2016.4218. PMID 27092831
- [Background] Winslow RL, Milligan ID, Voysey M, Luhn K, Shukarev G, Douoguih M, Snape MD. Immune Responses to Novel Adenovirus Type 26 and Modified Vaccinia Virus Ankara-Vectored Ebola Vaccines at 1 Year. JAMA. 2017 Mar 14;317(10):1075-1077. doi: 10.1001/jama.2016.20644. No abstract available. PMID 28291882
- See also: Oxford Vaccine Group homepage — http://www.ovg.ox.ac.uk/